CLINICAL TRIAL: NCT00632346
Title: Relationship of Adverse Childhood Experiences (Childhood Abuse, Neglect, and Household Dysfunction) to the Severity of Overweight and Obesity in Young Adults in a Military Dependent Population.
Brief Title: Relationship of Adverse Childhood Experiences to Overweight and Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Heather Elizondo Vega, CPT, USA, MC (Adolescent Medicine Fellow), Brooke Army Medical Center (U.S. Army)
Other Study IDs: C.2007.160
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Overweight; Obesity
Keywords: childhood abuse; overweight; obesity; BMI as a young adult; childhood physical abuse; childhood emotional abuse; childhood sexual abuse; childhood physical neglect; childhood emotional neglect; childhood witnessing of domestic violence; parental marital discord; household members with substance abuse; household members with mental illness; household members with criminal behavior; cumulative adverse childhood experiences
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 group: 200 patients presenting to the Adolescent Medicine Clinic at Brooke Army Medical Center between the ages of 18 and 23 years-old.

SUMMARY:
The purpose of this study is to determine if there is an association between a variety of adverse childhood experiences and overweight and obesity. The adverse childhood experiences that will be examined include childhood abuse (physical, emotional, sexual), childhood neglect (physical, emotional), and household dysfunction (domestic violence, parental marital discord, and household members with a history of substance abuse, mental illness, and criminal behavior). Because this study will be performed at a military treatment facility, additional military unique experiences to include frequent residential mobility and parental deployment will also be examined.

Hypotheses/Research Questions: Overweight and obese young adults are more likely to report having experienced adverse childhood experiences and household dysfunction than their peers of normal weight. In addition, the more severely overweight or obese the patient, the more likely the patient is to report a higher number of previous adverse childhood experiences. Thus, there is a graded relationship between the severity of overweight/obesity and the number of adverse childhood experiences.

DETAILED DESCRIPTION:
Previous studies have clearly demonstrated that there is an association between childhood adversities and a variety of eating and weight problems. The research can be extended by assessing the cumulative effects of adverse childhood experiences on the severity of overweight and obesity rather than focusing on individual categories of events. In addition, we can learn much by extending the research to include all overweight and obese patients, not just those who have a known underlying comorbid psychiatric disorder such as bulimia nervosa or binge eating disorder.

Lastly, the research on obesity and adverse childhood experiences should be extended to include younger subjects because obesity is now a public health problem of epidemic proportion in the United States, and it is now affecting younger and younger individuals.

The study proposed in this protocol will accomplish the goals of 1) assessing the cumulative effects of adverse childhood experiences, 2) assessing the association of these events with varying degrees of overweight and obesity, and 3) assessing this association in a younger population than that previously examined.

ELIGIBILITY:
Inclusion Criteria:

All patients presenting to the Adolescent Medicine clinic during the study period,

* both male and female,
* between the ages of 18 and 23 years of age,
* will be identified for possible participation in the study regardless of their health status, race, or body habitus.

Exclusion Criteria:

Only patients 18 years of age or older will be identified for possible participation in this study because such patients are not minors and could participate without parental consent.

* In addition, the questions from the questionnaire obtained from the Centers for Disease Control have only been assessed for reliability and validity in patients older than 18 years of age, and the questions are worded with the beginning phrase "During the first 18 years of life…"
* Lastly, requiring parental consent when inquiring about household dysfunction and a prior history of abuse would likely result in selection bias based on a higher number of subjects declining to participate. It is likely that more subjects will answer the questions truthfully if parental consent for participation is not required.
* Therefore, inclusion of younger patients would be a detriment to the scientific merit of the study, thus patients younger than age 18 will be excluded.
* The Brooke Army Medical Center Adolescent Medicine Clinic generally only serves patients 12-23 years of age. Therefore, patients above the age of 23 years will also be excluded.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female patients between the ages of 18 and 23 years of age who present to the Brooke Army Medical Center Adolescent Medicine Clinic(regardless of their gender, height, weight, blood pressure, reason for appointment, or health status)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Estimated); Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Relationship between reported prior Adverse Childhood Experiences (individual and cummulative) to weight status (underweight, normal weight, overweight, obese) in young adults (18-23 years-old) in a military dependent population. | BMI at one visit at the time of enrollment

SECONDARY OUTCOMES:
prevalence of underweight, normal weight, overweight, and obese in the population of 18-23 year-old military dependent patients | BMI at time of enrollment
prevalence of reported prior Adverse Childhood Experiences (individual and cummulative) reported by the population of 18-23 year-old military dependents | results of survey at time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Elizondo Vega, MD, Principal Investigator — U.S. Army, Brooke Army Medical Center, Adolescent Medicine Clinic, Department of Pediatrics
Locations (1):
- Adolescent Medicine Clinic, Brooke Army Medical Center, Fort Sam Houston, Texas, United States